CLINICAL TRIAL: NCT02889562
Title: Apixaban Versus Warfarin for the Management of Post-operative Atrial Fibrillation: a Prospective, Controlled, Randomized Pilot Study
Brief Title: Apixaban Versus Warfarin for the Management of Post-operative Atrial Fibrillation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sanford Health (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CV185-505
Record Dates: First submitted 2016-08-30; First posted 2016-09-05 (Estimated); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-12

CONDITIONS: Coronary Artery Bypass Grafting; Postoperative Atrial Fibrilation; Stroke; Systemic Embolism; Deep Venous Thrombosis
Keywords: apixaban; anticoagulant; CABG; thrombosis; fibrillation
MeSH Terms: conditions — Stroke; Venous Thrombosis; Thrombosis | interventions — apixaban; Warfarin

ARMS (2):
- Apixaban (Active Comparator): Apixaban is to be dosed at 5 mg by mouth twice daily, except in the case of the criteria listed below in "dose modifications". The duration of therapy will be at least 30 days. The patient's physician may determine that anticoagulation therapy should be continued after the study period, based on their examination of the patient at the 30-day post-operative examination.
  Interventions: Drug: Apixaban
- Warfarin (Active Comparator): While patients are hospitalized, warfarin will be dosed daily, with daily INR monitoring per hospital protocol. Daily doses may vary from 0.5mg to 15mg by mouth, as determined by patient specific factors such as patient size, hepatic function, INR, concomitant medications, diet, or other factors. Based on these factors or others not listed, there may also be days in which the patient is prescribed to not get does not receive a dose of warfarin.
  After discharge from the hospital, warfarin dosing will be subsequently managed by an anticoagulation clinic, per established protocols. All patients will have a goal INR of 2-3 during the duration of the study. The duration of therapy will be at least 30 days. The patient's physician may determine that anticoagulation therapy should be continued after the study period, based on their examination of the patient at the 30-day post-operative examination.
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Apixaban — Study arm that patient can be randomized to. Apixaban is a novel, orally active, potent, direct selective inhibitor of coagulation FXa that directly and reversibly binds to the active site of FXa and exerts anticoagulant and antithrombotic effects by diminishing the conversion of prothrombin to thrombin.
  Other Names: Eliquis
  Arms: Apixaban
Drug: Warfarin — Study arm that patient can be randomized to. Warfarin therapy has been the mainstay of therapy for patients with POAF. While the duration of therapy is usually short (3-4 weeks), complications of anticoagulation do occur. Additionally, warfarin therapy for POAF is associated with increased length of stay, need for monitoring, and bleeding complications.
  Other Names: Coumadin
  Arms: Warfarin

SUMMARY:
In this open-label, prospective, randomized pilot study, patients who develop atrial fibrillation after isolated coronary artery bypass grafting surgery will be identified. Patients with persistent atrial fibrillation (>12 hours) or recurrent sustained atrial fibrillation (>2 episodes of atrial fibrillation lasting longer than 30 minutes) will be candidates for inclusion. Upon meeting study inclusion and exclusion criteria, and after informed consent, patients will be randomized to either the standard of care (warfarin per protocol) or apixaban arms of the trial. Routine postoperative care after CABG will occur in both groups. Upon discharge, anticoagulation in both groups will be managed by the anticoagulation clinic. Patients will be followed for 30 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Signed Written Informed Consent
* Patients diagnosed with new-onset persistent or recurrent atrial fibrillation after isolated CABG surgery. Persistent atrial fibrillation is defined as an episode of >12 hours. Recurrent atrial fibrillation is defined as two or more episodes of atrial fibrillation lasting longer than 30 minutes.
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug. Patients undergoing isolated CABG must have this tested and documented prior to the procedure, and this will be verified prior to randomization.
* Women must not be breastfeeding.
* WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s): 30 days of treatment plus 5 half-lives of study drug Apixaban (3 days) or warfarin (8 days) plus 30 days (duration of ovulatory cycle) for a total of 38 days post-treatment completion.
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s): 30 days of treatment plus 5 half-lives of study drug Apixaban (3 days) or warfarin (8 days) plus 90 days (duration of sperm turnover) for a total of 98 days post-treatment completion.

Exclusion Criteria:

* Atrial fibrillation due to a reversible cause other than recent surgery
* Patients diagnosed with persistent or paroxysmal atrial fibrillation chronically before undergoing surgery
* Patients with mechanical heart valves
* Patients currently experiencing active bleeding precluding initialization of anticoagulation therapy in the opinion of their managing physician, or with increased bleeding risk (as determined by the attending surgeon) believed to be a contraindication to anticoagulation at the time of randomization Planned major surgery requiring stoppage of anticoagulation therapy during trial period
* Stroke within the previous 7 days
* Moderate or severe mitral stenosis
* Conditions other than atrial fibrillation that required anticoagulation (prosthetic mechanical heart valve)
* Patients taking warfarin, apixaban, rivaroxaban, dabigatran, edoxaban, clopidogrel, ticagrelor, or enoxaparin at home for any indication in the 15 days prior to surgery
* Patients requiring the use of clopidogrel or ticagrelor during the study period
* Severe renal insufficiency (serum creatinine level of >2.5 mg/dL or CrCL<25 ml/min) for consecutive measurements
* Allergies to warfarin or apixaban, or components of warfarin or apixaban

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-09; Primary Completion 2019-05-11 (Actual); Study Completion 2019-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelius Dyke, MD, Principal Investigator — Sanford Health
Locations (1):
- Sanford Health, Fargo, North Dakota, United States

REFERENCES:
- [Background] Anderson E, Johnke K, Leedahl D, Glogoza M, Newman R, Dyke C. Novel oral anticoagulants vs warfarin for the management of postoperative atrial fibrillation: clinical outcomes and cost analysis. Am J Surg. 2015 Dec;210(6):1095-102; discussion 1102-3. doi: 10.1016/j.amjsurg.2015.07.005. Epub 2015 Sep 18. PMID 26482512
- [Background] Schulman S, Angeras U, Bergqvist D, Eriksson B, Lassen MR, Fisher W; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in surgical patients. J Thromb Haemost. 2010 Jan;8(1):202-4. doi: 10.1111/j.1538-7836.2009.03678.x. Epub 2009 Oct 30. PMID 19878532
- [Background] Piccini JP, Zhao Y, Steinberg BA, He X, Mathew JP, Fullerton DA, Hegland DD, Hernandez AF, Mills RM, Klaskala W, Peterson ED. Comparative effectiveness of pharmacotherapies for prevention of atrial fibrillation following coronary artery bypass surgery. Am J Cardiol. 2013 Oct 1;112(7):954-60. doi: 10.1016/j.amjcard.2013.05.029. Epub 2013 Jul 11. PMID 23850476
- [Background] Lahiri MK, Fang K, Lamerato L, Khan AM, Schuger CD. Effect of race on the frequency of postoperative atrial fibrillation following coronary artery bypass grafting. Am J Cardiol. 2011 Feb 1;107(3):383-6. doi: 10.1016/j.amjcard.2010.09.032. PMID 21257002
- [Background] Rostagno C, La Meir M, Gelsomino S, Ghilli L, Rossi A, Carone E, Braconi L, Rosso G, Puggelli F, Mattesini A, Stefano PL, Padeletti L, Maessen J, Gensini GF. Atrial fibrillation after cardiac surgery: incidence, risk factors, and economic burden. J Cardiothorac Vasc Anesth. 2010 Dec;24(6):952-8. doi: 10.1053/j.jvca.2010.03.009. Epub 2010 May 31. PMID 20570180
- [Background] Raiten JM, Ghadimi K, Augoustides JG, Ramakrishna H, Patel PA, Weiss SJ, Gutsche JT. Atrial fibrillation after cardiac surgery: clinical update on mechanisms and prophylactic strategies. J Cardiothorac Vasc Anesth. 2015;29(3):806-16. doi: 10.1053/j.jvca.2015.01.001. No abstract available. PMID 26009291
- [Background] Fuster V, Ryden LE, Asinger RW, Cannom DS, Crijns HJ, Frye RL, Halperin JL, Kay GN, Klein WW, Levy S, McNamara RL, Prystowsky EN, Wann LS, Wyse DG, Gibbons RJ, Antman EM, Alpert JS, Faxon DP, Fuster V, Gregoratos G, Hiratzka LF, Jacobs AK, Russell RO, Smith SC Jr, Klein WW, Alonso-Garcia A, Blomstrom-Lundqvist C, de Backer G, Flather M, Hradec J, Oto A, Parkhomenko A, Silber S, Torbicki A; American College of Cardiology/American Heart Association Task Force on Practice Guidelines; European Society of Cardiology Committee for Practice Guidelines and Policy Conferences (Committee to Develop Guidelines for the Management of Patients With Atrial Fibrillation); North American Society of Pacing and Electrophysiology. ACC/AHA/ESC Guidelines for the Management of Patients With Atrial Fibrillation: Executive Summary A Report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the European Society of Cardiology Committee for Practice Guidelines and Policy Conferences (Committee to Develop Guidelines for the Management of Patients With Atrial Fibrillation) Developed in Collaboration With the North American Society of Pacing and Electrophysiology. Circulation. 2001 Oct 23;104(17):2118-50. No abstract available. PMID 11673357
- [Background] Granger CB, Alexander JH, McMurray JJ, Lopes RD, Hylek EM, Hanna M, Al-Khalidi HR, Ansell J, Atar D, Avezum A, Bahit MC, Diaz R, Easton JD, Ezekowitz JA, Flaker G, Garcia D, Geraldes M, Gersh BJ, Golitsyn S, Goto S, Hermosillo AG, Hohnloser SH, Horowitz J, Mohan P, Jansky P, Lewis BS, Lopez-Sendon JL, Pais P, Parkhomenko A, Verheugt FW, Zhu J, Wallentin L; ARISTOTLE Committees and Investigators. Apixaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2011 Sep 15;365(11):981-92. doi: 10.1056/NEJMoa1107039. Epub 2011 Aug 27. PMID 21870978
- [Background] Connolly SJ, Ezekowitz MD, Yusuf S, Eikelboom J, Oldgren J, Parekh A, Pogue J, Reilly PA, Themeles E, Varrone J, Wang S, Alings M, Xavier D, Zhu J, Diaz R, Lewis BS, Darius H, Diener HC, Joyner CD, Wallentin L; RE-LY Steering Committee and Investigators. Dabigatran versus warfarin in patients with atrial fibrillation. N Engl J Med. 2009 Sep 17;361(12):1139-51. doi: 10.1056/NEJMoa0905561. Epub 2009 Aug 30. PMID 19717844
- [Background] Patel MR, Mahaffey KW, Garg J, Pan G, Singer DE, Hacke W, Breithardt G, Halperin JL, Hankey GJ, Piccini JP, Becker RC, Nessel CC, Paolini JF, Berkowitz SD, Fox KA, Califf RM; ROCKET AF Investigators. Rivaroxaban versus warfarin in nonvalvular atrial fibrillation. N Engl J Med. 2011 Sep 8;365(10):883-91. doi: 10.1056/NEJMoa1009638. Epub 2011 Aug 10. PMID 21830957
- [Derived] Chapin TW, Leedahl DD, Brown AB, Pasek AM, Sand MG, Loy ML, Dyke CM. Comparison of Anticoagulants for Postoperative Atrial Fibrillation After Coronary Artery Bypass Grafting: A Pilot Study. J Cardiovasc Pharmacol Ther. 2020 Nov;25(6):523-530. doi: 10.1177/1074248420929483. Epub 2020 Jun 1. PMID 32476465
- See also: Apixaban. DrugPoints Summary. Micromedex 2.0. Truven Health Analytics, Inc. Greenwood Village, CO. — http://www.micromedexsolutions.com
- See also: Rivaroxaban. DrugPoints Summary. Micromedex 2.0. Truven Health Analytics, Inc. Greenwood Village, CO. — http://www.micromedexsolutions.com
- See also: Dabigatran Etexilate Mesylate. DrugPoints Summary. Micromedex 2.0. Truven Health Analytics, Inc. Greenwood Village, CO. — http://www.micromedexsolutions.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Warfarin: While patients are hospitalized, warfarin will be dosed daily, with daily INR monitoring per hospital protocol. Daily doses may vary from 0.5mg to 15mg by mouth, as determined by patient specific factors such as patient size, hepatic function, INR, concomitant medications, diet, or other factors. Based on these factors or others not listed, there may also be days in which the patient is prescribed to not get does not receive a dose of warfarin.
  After discharge from the hospital, warfarin dosing will be subsequently managed by an anticoagulation clinic, per established protocols. All patients will have a goal INR of 2-3 during the duration of the study. The duration of therapy will be at least 30 days. The patient's physician may determine that anticoagulation therapy should be continued after the study period, based on their examination of the patient at the 30-day post-operative examination.
  Warfarin: Study arm that patient can be randomized to. Warfarin therapy has been the mainstay of therapy for patients with POAF. While the duration of therapy is usually short (3-4 weeks), complications of anticoagulation do occur. Additionally, warfarin therapy for POAF is associated with increased length of stay, need for monitoring, and bleeding complications.
Period: Overall Study
Arm/Group | Apixaban | Warfarin
Started | 28 | 28
Completed | 28 | 26
Not Completed | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Apixaban | Warfarin | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.0 (8.1) | 69.5 (7.5) | 70.2 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 11
  Male | 25 | 20 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 28 | 27 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 28 | 56
Weight [Mean (Standard Deviation); unit: kg] | 98.6 (20.5) | 92.7 (17.2) | 95.6 (19.0)
Body Mass Index [Mean (Standard Deviation); unit: kg/meter-squared] | 32.4 (6.1) | 31.1 (5.6) | 31.7 (5.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Strokes
Description: Efficacy will be measured by the freedom from stroke during the study period. Events relating to stroke will be adjudicated using pre-determined definitions by independent committee members that remain blinded to the patient's treatment arm.
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 28 | 28
participants | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Apixaban vs Warfarin; Test type: Other — Pearson chi-squared tests or Fisher exact tests; p = 1.0, Chi-squared

2. Primary Outcome: Number of Participants With Thromboembolytic Events
Description: Efficacy will be measured by the freedom from thromboembolytic events during the study period. Events relating to thromboembolytic events will be adjudicated using pre-determined definitions by independent committee members that remain blinded to the patient's treatment arm.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 28 | 28
Participants | 0 | 0

3. Secondary Outcome: Units of Blood Given After Initiation of Anticoagulation Medication
Description: Units of blood or blood products given after the first dose of anticoagulation.
Time Frame: 30 days
Population: 2 units of blood were given per patient
Measure: Number; unit: total units of blood
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 28 | 28
total units of blood | 6 | 2

4. Secondary Outcome: Total Post-operative Length of Stay
Description: This will be measured from the date/time of the end of the subject's surgery until the date/time of the patient's discharge from the hospital. This will be measured in hours, to the nearest tenth of an hour.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 28 | 28
hours | 167.5 (76.6) | 143.1 (53.2)
Statistical Analysis 1: Comparison: Apixaban vs Warfarin; Test type: Other — t-test and Wilcoxon analysis; p = 0.17, t-test, 1 sided

5. Secondary Outcome: Time in Therapeutic Range of INR, if on Warfarin
Description: Time in therapeutic range of INR, if on warfarin, (eg. 2-3), measured as a percentage and defined for each patient using the Rosendaal equation
Time Frame: 30 days
Population: INR values are not measured for Apixaban. Apixaban is dose adjusted based on renal function, body weight, and age, but Warfarin requires laboratory monitoring due to other factors that may affect therapeutic affects such as prescribed and over-the-counter medications, consumption of alcoholic beverages, or a diet with inconsistent intake of vitamin K content.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 0 | 28
percentage |  | 56.8 (22.4)

ADVERSE EVENTS:
Time Frame: 30 days post-discharge, a total of up to 30 days
Arm/Group | Apixaban | Warfarin
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 1/28 | 1/28
Other Adverse Events (participants affected / at risk) | 14/28 | 7/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apixaban (N=28) | Warfarin (N=28)
required transfusions after discharge (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — received 2 units of blood
Subconjunctival hemorrhage (Eye disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apixaban (N=28) | Warfarin (N=28)
required transfusions after anticoagulation while in hospital (Blood and lymphatic system disorders) | 2 (2) | 1 (1) — 2 units of blood
GI bleed requiring endoscopy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epistaxis requiring intervention (Vascular disorders) | 2 (2) | 0 (0)
Epistaxis not requiring intervention (Vascular disorders) | 1 (1) | 0 (0)
Required thoracentesis (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 6 (6)

LIMITATIONS AND CAVEATS:
Limited by sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-05): https://cdn.clinicaltrials.gov/large-docs/62/NCT02889562/Prot_SAP_000.pdf